CLINICAL TRIAL: NCT04824664
Title: The ALIGHIERI Survey: an Italian Overview of Global Impact of tHe COVID-19 pandemIc on General surgERy practIce
Acronym: ALIGHIERI
Status: Completed | Type: Observational
Sponsor: Associazione Chirurghi Ospedalieri Italiani (Other)
Responsible Party: Principal Investigator, Pietro Fransvea, MD, Associazione Chirurghi Ospedalieri Italiani
Other Study IDs: Survey_ACOI_COVID19
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Surgery and covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — survey among surgeon

SUMMARY:
Introduction The present survey aimed to provide a comprehensive overview of the Italian scenario concerning general surgery during the first wave COVID-19 outbreak and evaluate the experiences, trends, attitudes, and possible educational outcomes that this emergency brought to light. Material and Methods A 31-item survey was designed and edited by the scientific board of the ACOI (Associazione Chirurghi Ospedalieri Italiani), addressing the impact of the pandemic outbreak on surgical staff and activity during the period from March 9 to May 30, 2020 (phase 1, lockdown period) and addressing the status of surgical activity, staff, and surgery resumption in the period from June 1 to September 30, 2020 (phase 3, restart). The survey was distributed via email and social media to Italian general surgeon working both in COVID-19 and non-COVID-19 hospitals. R

DETAILED DESCRIPTION:
Introduction The present survey aimed to provide a comprehensive overview of the Italian scenario concerning general surgery during the first wave COVID-19 outbreak and evaluate the experiences, trends, attitudes, and possible educational outcomes that this emergency brought to light. Material and Methods A 31-item survey was designed and edited by the scientific board of the ACOI (Associazione Chirurghi Ospedalieri Italiani), addressing the impact of the pandemic outbreak on surgical staff and activity during the period from March 9 to May 30, 2020 (phase 1, lockdown period) and addressing the status of surgical activity, staff, and surgery resumption in the period from June 1 to September 30, 2020 (phase 3, restart). The survey was distributed via email and social media to Italian general surgeon working both in COVID-19 and non-COVID-19 hospitals. .

ELIGIBILITY:
Inclusion Criteria:

* alla surgeon in activity

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all Italian general surgeon
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
surgery volume during covid19 lockdown | 8months
  number of surgical procedure performed all over italy during covid19 first lockdown

SECONDARY OUTCOMES:
surgery volume after the first covid19 lockdown | 3 months
  number of surgical procedure performed all over italy during re start period

CONTACTS AND LOCATIONS:
Locations (1):
- ACOI, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Cozza V, Fransvea P, La Greca A, De Paolis P, Marini P, Zago M, Sganga G; I.-ACTSS.-COVID19 Collaborative Study Group. I-ACTSS-COVID-19-the Italian acute care and trauma surgery survey for COVID-19 pandemic outbreak. Updates Surg. 2020 Jun;72(2):297-304. doi: 10.1007/s13304-020-00832-4. Epub 2020 Jun 24. PMID 32583216
- [Result] Fransvea P, Sganga G, Cozza V, Di Grezia M, Fico V, Tirelli F, Pepe G, La Greca A. Set up of a dedicated COVID-19 surgical pathway and operating room for surgical emergencies. J Trauma Acute Care Surg. 2020 Oct;89(4):e97-e100. doi: 10.1097/TA.0000000000002852. No abstract available. PMID 33017138